CLINICAL TRIAL: NCT07290725
Title: Cross-cultural Adaptation and Translation Validation of the iADH Universal Case Mix Tool (UCMT).
Acronym: CCV UCMT
Status: Enrolling by invitation | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Collaborators: University of Freiburg (Other); Universidad Catolica de Cordoba (Unknown); University of Chile (Other)
Responsible Party: Principal Investigator, Sebastian Veliz, DDS, Researcher, Sigmund Freud PrivatUniversitat
Other Study IDs: 17793138
Record Dates: First submitted 2025-11-26; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dentistry
Keywords: special care dentistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- special care dentists - spanish: Special Care Dentistry Specialist, native Spanish speaker
- Special care dentists - german: Special Care Dentistry Specialist, native German speaker
- Special care dentists - Portuguese: Special Care Dentistry Specialist, native Portuguese speaker

SUMMARY:
This study aims to translate, culturally adapt, and validate the iADH Universal Case Mix Tool (UCMT) for dental care professionals working with people with disabilities.

The study will assess linguistic accuracy, applicability, and reliability/validity of the German, Spanish and Portuguese version of the instrument.

DETAILED DESCRIPTION:
This study is a multicentre, non-interventional methodological study aimed at translating, culturally adapting, and validating the iADH Universal case mix tool (UCMT) for use by dental care professionals working with people living with disabilities; following international guidelines for cross-cultural adaptation of measurement instruments.

The translation and cultural adaptation process will include forward and backward translations of the original UCMT (English) to German, Spanish and Portuguese. Two independent forward translations will be performed for each language, followed by reconciliation into a single version, based on semantic equivalence, clarity and cultural appropriatness. Blinded backward translations into English will then be conducted to ensure conceptual consistency with the original instrument.

A panel of experts, composed of dental experts and linguistic professionals fluent in both languages will review all trnaslated versions using a Delphi approach.Later, the adapted instruments will be reviewed by the original UCMT developers for the final approval. Concent Validity Index (CVI) of the translated UCMT will be evaluated through expert ratings and cognitive interviews with dental professionals experienced in special care dentistry.

Following the experts' validation, a pilot reliability phase will be conducted using standarised online clinical cases developed for the original versions of the UCMT. Participating raters will complete a online questionnaire using the translated UCMT. Intra and interrater agreement will be assessed to evaluate consistency of the translated instrument in a simulated clinical scenario.

This study does not involve real patients of the collection of sensitive personal data.

ELIGIBILITY:
Inclusion Criteria:

* Special care dentist
* Native in German, Spanish or Portuguese
* Agree to participate, complete the instrument 2 times

Exclusion Criteria:

* Not meeting the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * Special care dentist
  * Native in German, Spanish or Portuguese
  * Agree to participate, complete the instrument 2 times
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Content validity of the translated UCMT | 1 week
  Content validity of the UCMT will be assessed by a panel of multidisciplinary experts, assessing clarity, relevance and cultural appropiatness. Experts ratings will be used to calculate Content Validity Index (CVI) for the translated versions of the UCMT.
  Unit of measure: CVI (Range 0-1)

SECONDARY OUTCOMES:
Interrater agreement of the UCMT domains scores | 1 month
  Interrater agreement will be assesed based on scores asigned to the seven domains of the UCMT in the original version and validation. Raters will independently evaluate standarised online cases using the translated versions of the UCMT. Agreement between raters will be quantified for each UCMT domain.
  Unit of measure:
  Interclass correlation coeficiente (range 0-1)
Temporal stability (Test-retest) of UCMT domain scores | 2 weeks
  intrarater agreement (Temporal stability) will be assesed based on scores asigned to the seven domains of the UCMT in the original version and validation. Raters will independently evaluate standarised online cases using the translated versions of the UCMT on two occasiions separated by 1-2 weeks . Agreement between these occasions will be quantified for each UCMT domain.
  Unit of measure:
  Interclass correlation coeficiente (range 0-1)

CONTACTS AND LOCATIONS:
Locations (1):
- SFU - Online questionnaire, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Not necessary

REFERENCES:
- [Background] Mac Giolla Phadraig C, Faulks D, McGrath C, Dougall A, Molina G. Development and Content Validity of the International Association for Disability and Oral Health Universal Case Mix Tool: A Consensus Study. Community Dent Oral Epidemiol. 2025 Aug;53(4):402-412. doi: 10.1111/cdoe.13041. Epub 2025 Apr 30. PMID 40304234